CLINICAL TRIAL: NCT03611530
Title: Randomized, Double-blind, Controlled Trial Evaluating the Effects of an Ophthalmic Solution of Coenzyme Q10 and Vitamin E in Patients Affected by Open-angle Glaucoma
Brief Title: CoQun Study - (COQUN): a Study to Evaluate the Effects of CoQun in Patients Affected by Open-angle Glaucoma
Acronym: CoQun
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRFMN-OG-7204
Record Dates: First submitted 2017-09-04; First posted 2018-08-02 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Prostaglandins, Synthetic; Prostaglandins A

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CoQun® (Experimental): Patients in Arm A will be randomized to receive Prostaglandin analogue (PGA) monotherapy + CoQun®. CoQun® ophthalmic solution will be administered two times daily. CoQun® will be administered in addition to hypotensive therapy. Dose modifications for CoQun® are not permitted.
  Interventions: Device: Coqun® ophthalmic solution
- Placebo (Placebo Comparator): Patients in Arm B will be randomized to receive Prostaglandin analogue (PGA) monotherapy +Placebo. Placebo ophthalmic solution will be administered two times daily. Placebo will be administered in addition to hypotensive therapy. Dose modifications for Placebo are not permitted.
  Interventions: Other: Placebo ophthalmic solution

INTERVENTIONS:
Device: Coqun® ophthalmic solution — Prostaglandin analogue (PGA) monotherapy + Coqun® ophthalmic solution
  Other Names: Prostaglandin analogue (PGA) monotherapy
  Arms: CoQun®
Other: Placebo ophthalmic solution — Prostaglandin analogue (PGA) monotherapy + Placebo ophthalmic solution
  Other Names: Prostaglandin analogue (PGA) monotherapy
  Arms: Placebo

SUMMARY:
This is a randomized, parallel arm, multicenter, double-blind trial.

Patients with POAG will be randomized 1:1 ratio to receive:

* Prostaglandin analogue (PGA) monotherapy + CoQun® (Arm A)
* Prostaglandin analogue (PGA) monotherapy + Vehicle (Arm B)

DETAILED DESCRIPTION:
CoQun® 10 ml is a medical device marked by the European Community as class IIb. This device has a system of dispensation that permits it to be preservative free (OSD - Ophthalmic Squeeze Dispenser). Investigators and patients will be masked to the study treatment. In order to mask the treatment, identical kit boxes, identical packaging (bottles and labels) will be used for vehicle and active product. The bottles will be dispensed sealed to the patient.

One or two drops of the solution (CoQun® or Vehicle) will be instilled in the conjunctival sac of both eyes, twice daily from 8 to 10 AM and from 8 to 10 PM. Hypotensive therapy should be administered in the evening one hour after the CoQun® or Vehicle administration.

At baseline, ocular hypotensive treatment, as per inclusion criteria has to be a PGA monotherapy. During the follow-up, in case the IOP exceeds 28 mmHg, any additional hypotensive therapy will be allowed to obtain IOP control.

Dose modifications/reductions of CoQun® /Vehicle are not permitted.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosis of POAG (monolateral or bilateral) with an IOP ranging from 17 to 21 mm Hg (at the last performed visit and confirmed at the baseline study visit) on treatment with a topical prostaglandin analogue (PGA) monotherapy.
2. VF examination at randomization: VF Mean Defect (MD) at baseline within -4 decibel (dB) and -10dB and VF Pattern Standard Deviation (PSD) within 4 dB and 10dB (stage 2-3 per the Enhanced Glaucoma Staging System 2 (GSS) determined by Humphrey Field Analyzer II-i, program 30-2 SITA standard.
3. In order to determine patient's reliability to perform VF examination: before baseline VF, at least two reliable VF examinations during the last year had to be performed. Visual fields are considered reliable if false-positive responses are fewer than 15% and a clear blind spot could be seen in the VF printouts, threshold value <10 dB.
4. Age >40 years
5. Provision of informed consent prior to any study specific procedures

Exclusion Criteria:

1. Secondary glaucoma (exofoliative glaucoma, pigmentary glaucoma, neovascular glaucoma).
2. Abnormalities of the anterior segment of the eye that could affect IOP assessment.
3. Cornea abnormalities with entities that could affect IOP evaluation.
4. Other conditions different from glaucoma that could cause VF abnormalities (degenerative myopia, diabetic retinopathy, maculopathy, other optic nerve abnormalities that could mimic glaucoma damage).
5. BCVA) < 0.5 Snellen decimal fraction
6. Any previous ocular surgery except for uncomplicated cataract extraction and YAG laser capsulotomy, laser glaucoma surgeries (argon laser trabeculoplasty and/or selective laser trabeculoplasty).
7. Pregnancy or breast-feeding.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Time to Progression (TTP) | Randomization till VF progression, up to 36 months
  Time to Progression (TTP) defined as the time between baseline visit and the visit with the first evidence of progression in either eye is detected. When progression is detected, the progression should be confirmed at the two subsequent and consecutive Visual Field (VF) examinations.VF examinations will be assessed by an independent reading centre.

SECONDARY OUTCOMES:
Velocity of Visual Field (VF) loss | Randomization till VF progression, up to 36 months
  VF loss as determined by Guided Progression Analysis software (version 5.1.1) will be assessed at the last VF examination.
Retinal Nerve Fiber Layer (RNFL) thickness | Randomization till VF progression, up to 36 months
  RNFL thickness by the means of OCT: change from baseline
Intraocular pressure (IOP) | Randomization till VF progression, up to 36 months
  IOP change from baseline
Best Correct Visual Acuity (BCVA) | Randomization till VF progression, up to 36 months
  BCVA change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Quaranta, MD PhD, Principal Investigator — Università degli Studi di Brescia
Locations (1):
- Università degli Studi di Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quaranta L, Riva I, Biagioli E, Rulli E, Rulli E, Poli D, Legramandi L; CoQun(R) Study Group. Evaluating the Effects of an Ophthalmic Solution of Coenzyme Q10 and Vitamin E in Open-Angle Glaucoma Patients: A Study Protocol. Adv Ther. 2019 Sep;36(9):2506-2514. doi: 10.1007/s12325-019-01023-3. Epub 2019 Jul 12. PMID 31301054